CLINICAL TRIAL: NCT02498860
Title: Efficacy and Safety of Pemetrexed Plus Cisplatin as Combination Chemotherapy for Post-operative Adenocarcinoma : Multi-center, Single Arm, Open-label, Phase Ⅱ Trial
Brief Title: Efficacy and Safety of Adjuvant Pemetrexed Plus Cisplatin for Adenocarcinoma of Lung
Acronym: APICAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Kosin University Gospel Hospital (Other); Korea University Guro Hospital (Other); Severance Hospital (Other); Chungnam National University Hospital (Other); Kyungpook National University Hospital (Other); Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNUHH-2015-7
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Adenocarcinoma; Lung Neoplasm
Keywords: adenocarcinoma; lung; adjuvant chemotherapy; pemetrexed; cisplatin; surgery
MeSH Terms: conditions — Adenocarcinoma; Lung Neoplasms | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemebit plus Cisplatin (Experimental): Pemetrexed (Pemebit 500 mg/m2) plus cisplatin (75 mg/m2) every 3 weeks up to 4 cycles
  Interventions: Drug: Pemebit; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemebit — 500mg/m2 on day 1 of every 3-week cycle, for a maximum of 4 cycles
  Other Names: Pemetrexed
Drug: Cisplatin — 75mg/m2 on day 1 of every 3-week cycle, for a maximum of 4 cycles

SUMMARY:
Two-Year Disease Free Survival Rate of Stage IB~IIIA adenocarcinoma after Adjuvant Chemotherapy with Pemetrexed and Cisplatin will be assessed. A total of 106 patients will be recruited for 12 months, and followed for two years, thus the duration of study will be 36 months.

DETAILED DESCRIPTION:
Primary endpoint : 2 year disease free survival

Secondary endpoints:

Overall survival, Frequency and severity of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of Lung
* Postoperative pathologic stage IB~IIIA
* Complete surgical resection (R0 resection) N1-2: R0 resection with lobectomy and mediastinal lymph nodes dissection (MLND) N0: R0 resection with lobectomy with or without MLND
* Adjuvant treatment should start between 4 to 6 weeks after surgery
* ECOG performance status 0-1
* Weight loss during last 3 months should be less than 10%.
* Normal hematologic, hepatic and renal function Neutrophil count > 1500 /microliter, Platelet > 100,000/microliter, Hemoglobin > 9 g/dL Bilirubin <=1.5 x upper limit normal, transaminase < 2.5 x upper limit normal Serum Creatinine <=1.5 mg/dL
* Women in child bearing age should consent using contraceptive measures, and must have negative pregnancy test.

Exclusion Criteria:

* Other malignant neoplastic disease within 5 years.
* Neoadjuvant chemotherapy before surgery of lung cancer
* Patients who will be treated with postoperative radiation.
* Stage IIIB or IV lung cancer
* Severe infection, or cardiorespiratory, hematologic illness
* HIV positive cases
* Pregnancy or lactating women
* Autoimmune diseases or those who receiving immune suppressive treatment
* Symptomatic neuropathy > CTCAE grade 1
* Those who consented other clinical trials within 3 months
* Other significant medical conditions contraindicated to clinical trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Disease free survival rate | 2 year
  Disease free survival time is measured from the date of enrollment to date of tumor recurrence.

SECONDARY OUTCOMES:
Overall survival | 4 year
  Overall survival time is measured from the date of enrollment to date of death from any cause. Participants who are alive when the data lock or is lost to follow-up will have their overall survival time censored on the last date the participant is known to be alive.
Adverse events | 4 months
  adverse events using common terminology criteria for adverse events 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Study Chair — Chonnam National University Hospital
Locations (7):
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Kyungpook National University Medical Center, Daegu, Kyungpook
  - Chungnam National University Hospital, Daejeon
  - Pusan National University Hospital, Pusan
  - Kosin University Gospel Hospital, Pusan
  - Korea university Guro hospital, Seoul
  - Severance hospital, Seoul

REFERENCES:
- [Result] Kreuter M, Vansteenkiste J, Fischer JR, Eberhardt W, Zabeck H, Kollmeier J, Serke M, Frickhofen N, Reck M, Engel-Riedel W, Neumann S, Thomeer M, Schumann C, De Leyn P, Graeter T, Stamatis G, Zuna I, Griesinger F, Thomas M; TREAT investigators. Randomized phase 2 trial on refinement of early-stage NSCLC adjuvant chemotherapy with cisplatin and pemetrexed versus cisplatin and vinorelbine: the TREAT study. Ann Oncol. 2013 Apr;24(4):986-92. doi: 10.1093/annonc/mds578. Epub 2012 Nov 15. PMID 23161898
- [Result] Douillard JY, Rosell R, De Lena M, Carpagnano F, Ramlau R, Gonzales-Larriba JL, Grodzki T, Pereira JR, Le Groumellec A, Lorusso V, Clary C, Torres AJ, Dahabreh J, Souquet PJ, Astudillo J, Fournel P, Artal-Cortes A, Jassem J, Koubkova L, His P, Riggi M, Hurteloup P. Adjuvant vinorelbine plus cisplatin versus observation in patients with completely resected stage IB-IIIA non-small-cell lung cancer (Adjuvant Navelbine International Trialist Association [ANITA]): a randomised controlled trial. Lancet Oncol. 2006 Sep;7(9):719-27. doi: 10.1016/S1470-2045(06)70804-X. PMID 16945766
- [Result] Olaussen KA, Dunant A, Fouret P, Brambilla E, Andre F, Haddad V, Taranchon E, Filipits M, Pirker R, Popper HH, Stahel R, Sabatier L, Pignon JP, Tursz T, Le Chevalier T, Soria JC; IALT Bio Investigators. DNA repair by ERCC1 in non-small-cell lung cancer and cisplatin-based adjuvant chemotherapy. N Engl J Med. 2006 Sep 7;355(10):983-91. doi: 10.1056/NEJMoa060570. PMID 16957145
- [Derived] Park CK, Oh HJ, Yoo SS, Lee SY, Lee SH, Kim EY, Lee SY, Choi J, Lee MK, Kim MH, Jang TW, Chung C, Oh IJ, Kim YC. Open-label, multi-center, phase II study of adjuvant pemetrexed plus cisplatin for completely resected stage IB to IIIA adenocarcinoma of the lung: APICAL trial. Transl Lung Cancer Res. 2022 Aug;11(8):1606-1618. doi: 10.21037/tlcr-22-183. PMID 36090637